CLINICAL TRIAL: NCT04528173
Title: Opioid-Free Versus Transitional Anesthetic With Opioids From Tonsillectomy
Brief Title: Opioid-Free Anesthetic for Tonsillectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other); University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-016618
Record Dates: First submitted 2020-07-28; First posted 2020-08-27 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia; Opioid Use; Tonsillitis; Sleep Disorder; Surgery
Keywords: Tonsillectomy; Opioid-Free; Ketorolac; Dexmedetomidine; Acute postoperative pain relief; Opioid; Morphine; Fentanyl
MeSH Terms: conditions — Tonsillitis; Sleep Wake Disorders | interventions — Ketorolac; Ketorolac Tromethamine; Dexmedetomidine; Morphine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Subject will be randomized to 1:1 intra-operative opioid-free (OFG) vs traditional care anesthetic with opioids (TCG) group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The unblinded members are the treating anesthesiologist for the case, staff who randomize, and collect and enter intra-op medications into electronic data capture (EDC).
  Blinded members include the subject/family members, the surgeon, staff who perform post-op assessment, physician investigator who perform any adverse event/serious adverse event (AE/SAE) assessments, statistician and data safety monitoring board (DSMB).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Traditional Care Group (TCG) (Active Comparator): Traditional anesthetic with opioids group will receive institutional standard clinical care for tonsillectomy, including a standardized opioid dose at the beginning of the case and again at the end if needed. Dexmedetomidine and Ketorolac will not be used intra-operatively in this cohort to prevent confounding.
  Interventions: Drug: Morphine; Drug: Fentanyl
- Opioid-Free Group (OFG) (Experimental): Opioid-Free group will receive institutional standard clinical care for tonsillectomy, without opioids, but including Dexmedetomidine and Ketorolac.
  Interventions: Drug: Ketorolac; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketorolac — Ketorolac (0.5mg/kg; maximum 15mg intravenously) will be given at end of procedure after evaluation for hemostasis.
  Other Names: Toradol
  Arms: Opioid-Free Group (OFG)
Drug: Dexmedetomidine — Dexmedetomidine (1ug/kg with maximum 50ug intravenously) will be given at beginning of procedure.
  Other Names: Precedex
  Arms: Opioid-Free Group (OFG)
Drug: Morphine — Morphine (0.05-0.1 mg/kg intravenously) will be given intra-operatively per institutional standard clinical care.
  Arms: Traditional Care Group (TCG)
Drug: Fentanyl — Fentanyl (0.5-2 ug/kg intravenously) will be given intra-operatively per institutional standard clinical care.
  Arms: Traditional Care Group (TCG)

SUMMARY:
Prospective randomized controlled trial to determine if opioid-free anesthetic for tonsillectomy is non-inferior to standard opioid-containing anesthetic

DETAILED DESCRIPTION:
Objectives:

Primary: To determine if an opioid-free anesthetic provides equivalent acute postoperative pain relief in tonsillectomy.

Secondary: To determine if post-operative pain at home is not significantly different with an opioid-free regimen compared to an opioid containing regimen for tonsillectomy.

Study Design: Prospective, randomized, multi-center trial study

Study Interventions and Measures:

Subject will be randomized to 1:1 intra-operative opioid-free (OFG) vs traditional care anesthetic with opioids (TCG) group

The primary endpoint is the median pain score (calculated by a blinded validated observer in the recovery room at two time intervals) between the two cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 2 to 18 years.
2. American Society of Anesthesiologists {ASA) ≤ 3 physical classification system
3. Girls after menarche must have a negative pregnancy test.
4. Scheduled tonsillectomy or tonsillectomy combined with adenoidectomy and/or ear tube placement at the Children's Hospital of Philadelphia (CHOP) main or ambulatory surgical centers.
5. Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

1. Current (Within the last 30 days) opioid use for pain control
2. High risk for surgical site hemorrhage, determined by bleeding disorder diagnosis or evidence or poor hemostasis
3. Multiple scheduled surgeries at the same time other than adenoidectomy and/or ear tube placement
4. History of drug abuse, chronic pain, bleeding disorder
5. Chronic disease such as sickle cell disease for which treatment with opioids may be clinically indicated
6. Significant congenital disorders, medication allergies or comorbidities, specifically a pre-disposition to bradycardia or conduction abnormalities, cyanotic cardiac disease and use of medications that would increase risk of bleeding or bradycardia.
7. History of hepatic dysfunction, renal dysfunction, thrombocytopenia, or anemia (including pre-surgery laboratory abnormalities)
8. History of hypersensitivity to NSAIDs
9. Patients with asthma, including patients who have experienced aspirin- or NSAID-sensitive asthma or a history of exacerbation when aspirin or NSAIDs are administered (e.g. bronchospasm, urticaria, etc.)
10. Subjects receiving medications that could impact metabolism of either study drug should also be excluded
11. Trisomy 21 diagnosis
12. Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.
13. Patients on a Ketogenic diet
14. Parents or subjects who do not speak English

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tori Sutherland, MD,MPH, Principal Investigator — Children's Hospital of Philadelphia; Anthony Sheyn, MD, FACS, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center; St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- [Background] Volkow ND, Jones EB, Einstein EB, Wargo EM. Prevention and Treatment of Opioid Misuse and Addiction: A Review. JAMA Psychiatry. 2019 Feb 1;76(2):208-216. doi: 10.1001/jamapsychiatry.2018.3126. PMID 30516809
- [Background] Scholl L, Seth P, Kariisa M, Wilson N, Baldwin G. Drug and Opioid-Involved Overdose Deaths - United States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2018 Jan 4;67(5152):1419-1427. doi: 10.15585/mmwr.mm675152e1. PMID 30605448
- [Background] Harbaugh CM, Lee JS, Hu HM, McCabe SE, Voepel-Lewis T, Englesbe MJ, Brummett CM, Waljee JF. Persistent Opioid Use Among Pediatric Patients After Surgery. Pediatrics. 2018 Jan;141(1):e20172439. doi: 10.1542/peds.2017-2439. Epub 2017 Dec 4. PMID 29203521
- [Background] Harbaugh CM, Nalliah RP, Hu HM, Englesbe MJ, Waljee JF, Brummett CM. Persistent Opioid Use After Wisdom Tooth Extraction. JAMA. 2018 Aug 7;320(5):504-506. doi: 10.1001/jama.2018.9023. PMID 30088000
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Background] Franz AM, Dahl JP, Huang H, Verma ST, Martin LD, Martin LD, Low DK. The development of an opioid sparing anesthesia protocol for pediatric ambulatory tonsillectomy and adenotonsillectomy surgery-A quality improvement project. Paediatr Anaesth. 2019 Jul;29(7):682-689. doi: 10.1111/pan.13662. Epub 2019 Jun 19. PMID 31077491
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933
- [Background] Elkassabany NM, Mariano ER. Opioid-free anaesthesia - what would Inigo Montoya say? Anaesthesia. 2019 May;74(5):560-563. doi: 10.1111/anae.14611. Epub 2019 Feb 25. No abstract available. PMID 30802930
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update). Otolaryngol Head Neck Surg. 2019 Feb;160(1_suppl):S1-S42. doi: 10.1177/0194599818801757. PMID 30798778
- [Background] Baugh RF, Archer SM, Mitchell RB, Rosenfeld RM, Amin R, Burns JJ, Darrow DH, Giordano T, Litman RS, Li KK, Mannix ME, Schwartz RH, Setzen G, Wald ER, Wall E, Sandberg G, Patel MM; American Academy of Otolaryngology-Head and Neck Surgery Foundation. Clinical practice guideline: tonsillectomy in children. Otolaryngol Head Neck Surg. 2011 Jan;144(1 Suppl):S1-30. doi: 10.1177/0194599810389949. PMID 21493257
- [Background] Cote CJ, Posner KL, Domino KB. Death or neurologic injury after tonsillectomy in children with a focus on obstructive sleep apnea: houston, we have a problem! Anesth Analg. 2014 Jun;118(6):1276-83. doi: 10.1213/ANE.0b013e318294fc47. PMID 23842193
- [Background] McCabe SE, Schulenberg JE, O'Malley PM, Patrick ME, Kloska DD. Non-medical use of prescription opioids during the transition to adulthood: a multi-cohort national longitudinal study. Addiction. 2014 Jan;109(1):102-10. doi: 10.1111/add.12347. Epub 2013 Oct 22. PMID 24025114
- [Background] McCabe SE, West BT, Boyd CJ. Medical use, medical misuse, and nonmedical use of prescription opioids: results from a longitudinal study. Pain. 2013 May;154(5):708-713. doi: 10.1016/j.pain.2013.01.011. Epub 2013 Jan 26. PMID 23433943
- [Background] McCabe SE, West BT, Boyd CJ. Leftover prescription opioids and nonmedical use among high school seniors: a multi-cohort national study. J Adolesc Health. 2013 Apr;52(4):480-5. doi: 10.1016/j.jadohealth.2012.08.007. Epub 2012 Nov 22. PMID 23298996
- [Background] Winters KC, Arria A. Adolescent Brain Development and Drugs. Prev Res. 2011;18(2):21-24. PMID 22822298
- [Background] Mason KP. Paediatric emergence delirium: a comprehensive review and interpretation of the literature. Br J Anaesth. 2017 Mar 1;118(3):335-343. doi: 10.1093/bja/aew477. PMID 28203739
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Althunian TA, de Boer A, Klungel OH, Insani WN, Groenwold RH. Methods of defining the non-inferiority margin in randomized, double-blind controlled trials: a systematic review. Trials. 2017 Mar 7;18(1):107. doi: 10.1186/s13063-017-1859-x. PMID 28270184
- [Background] Strom BL, Berlin JA, Kinman JL, Spitz PW, Hennessy S, Feldman H, Kimmel S, Carson JL. Parenteral ketorolac and risk of gastrointestinal and operative site bleeding. A postmarketing surveillance study. JAMA. 1996 Feb 7;275(5):376-82. PMID 8569017
- [Background] Forrest JB, Camu F, Greer IA, Kehlet H, Abdalla M, Bonnet F, Ebrahim S, Escolar G, Jage J, Pocock S, Velo G, Langman MJ, Bianchi PG, Samama MM, Heitlinger E; POINT Investigators. Ketorolac, diclofenac, and ketoprofen are equally safe for pain relief after major surgery. Br J Anaesth. 2002 Feb;88(2):227-33. doi: 10.1093/bja/88.2.227. PMID 11883386
- [Background] Mowatt G, Cook JA, Fraser C, McKerrow WS, Burr JM. Systematic review of the safety of electrosurgery for tonsillectomy. Clin Otolaryngol. 2006 Apr;31(2):95-102. doi: 10.1111/j.1749-4486.2006.01162.x. PMID 16620327
- [Background] Chan DK, Parikh SR. Perioperative ketorolac increases post-tonsillectomy hemorrhage in adults but not children. Laryngoscope. 2014 Aug;124(8):1789-93. doi: 10.1002/lary.24555. Epub 2014 May 27. PMID 24338331
- [Background] McClain K, Williams AM, Yaremchuk K. Ketorolac usage in tonsillectomy and uvulopalatopharyngoplasty patients. Laryngoscope. 2020 Apr;130(4):876-879. doi: 10.1002/lary.28077. Epub 2019 May 30. PMID 31145482
- [Background] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Background] Olutoye OA, Glover CD, Diefenderfer JW, McGilberry M, Wyatt MM, Larrier DR, Friedman EM, Watcha MF. The effect of intraoperative dexmedetomidine on postoperative analgesia and sedation in pediatric patients undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Aug;111(2):490-5. doi: 10.1213/ANE.0b013e3181e33429. Epub 2010 Jul 7. PMID 20610555
- [Background] Lee MS, Montague ML, Hussain SS. Post-tonsillectomy hemorrhage: cold versus hot dissection. Otolaryngol Head Neck Surg. 2004 Dec;131(6):833-6. doi: 10.1016/j.otohns.2004.08.008. PMID 15577776
- [Background] Diercks GR, Comins J, Bennett K, Gallagher TQ, Brigger M, Boseley M, Gaudreau P, Rogers D, Setlur J, Keamy D, Cohen MS, Hartnick C. Comparison of Ibuprofen vs Acetaminophen and Severe Bleeding Risk After Pediatric Tonsillectomy: A Noninferiority Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2019 Jun 1;145(6):494-500. doi: 10.1001/jamaoto.2019.0269. PMID 30946442
- [Background] Mroszczak EJ, Jung D, Yee J, Bynum L, Sevelius H, Massey I. Ketorolac tromethamine pharmacokinetics and metabolism after intravenous, intramuscular, and oral administration in humans and animals. Pharmacotherapy. 1990;10(6 ( Pt 2)):33S-39S. PMID 2082311
- [Background] Macario A, Lipman AG. Ketorolac in the era of cyclo-oxygenase-2 selective nonsteroidal anti-inflammatory drugs: a systematic review of efficacy, side effects, and regulatory issues. Pain Med. 2001 Dec;2(4):336-51. doi: 10.1046/j.1526-4637.2001.01043.x. PMID 15102238
- [Background] Mitchell RB, Archer SM, Ishman SL, Rosenfeld RM, Coles S, Finestone SA, Friedman NR, Giordano T, Hildrew DM, Kim TW, Lloyd RM, Parikh SR, Shulman ST, Walner DL, Walsh SA, Nnacheta LC. Clinical Practice Guideline: Tonsillectomy in Children (Update)-Executive Summary. Otolaryngol Head Neck Surg. 2019 Feb;160(2):187-205. doi: 10.1177/0194599818807917. PMID 30921525
- [Background] Mudd PA, Thottathil P, Giordano T, Wetmore RF, Elden L, Jawad AF, Ahumada L, Galvez JA. Association Between Ibuprofen Use and Severity of Surgically Managed Posttonsillectomy Hemorrhage. JAMA Otolaryngol Head Neck Surg. 2017 Jul 1;143(7):712-717. doi: 10.1001/jamaoto.2016.3839. PMID 28472239
- [Background] Gupta P, Whiteside W, Sabati A, Tesoro TM, Gossett JM, Tobias JD, Roth SJ. Safety and efficacy of prolonged dexmedetomidine use in critically ill children with heart disease*. Pediatr Crit Care Med. 2012 Nov;13(6):660-6. doi: 10.1097/PCC.0b013e318253c7f1. PMID 22791093
- [Background] Mahmoud M, Mason KP. Dexmedetomidine: review, update, and future considerations of paediatric perioperative and periprocedural applications and limitations. Br J Anaesth. 2015 Aug;115(2):171-82. doi: 10.1093/bja/aev226. PMID 26170346
- [Background] Tsiotou AG, Malisiova A, Kouptsova E, Mavri M, Anagnostopoulou M, Kalliardou E. Dexmedetomidine for the reduction of emergence delirium in children undergoing tonsillectomy with propofol anesthesia: A double-blind, randomized study. Paediatr Anaesth. 2018 Jul;28(7):632-638. doi: 10.1111/pan.13397. Epub 2018 May 12. PMID 29752853
- See also: Key substance use and mental health indicators in the United States: Results from the 2016 National Survey on Drug Use and Health (HHS Publication No. SMA 17-5044). Center f — https://www.samhsa.gov/data/
- See also: Sealed Envelope Ltd. 2012. Power calculator for continuous outcome non-inferiority trial. — https://www.sealedenvelope.com/power/continuous-noninferior/
- See also: Buck, ML. Use of Intravenous Ketorolac for Postoperative Analgesia in Infants: Pediatric Pharmacotherapy, A Monthly Newsletter. . 2011 — https://med.virginia.edu/pediatrics/wp-content/uploads/sites/237/2015/12/201108.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG) | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Customized [Mean (Full Range); unit: years] | 3.56 [2 to 7] | 6.47 [3 to 13] | 4.97 [2 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean FLACC (Face, Legs, Activity, Cry, Consolability) Pain Score
Description: Mean FLACC pain assessment scores are calculated 15 and 30 minutes after awakening, Scores are calculated by a blinded study team observer. Minimum Score: 0 and Maximum Score: 10. Higher scores indicate worse outcomes.
  One Nursing Maximum FLACC pain score is obtained by an unblinded patient Registered Nurse (RN) during the patient's Post-Anesthesia Care Unit (PACU) stay within one hour of awakening. The pain score is collected from the nursing documentation in the electronic medical record. FLACC Minimum Score: 0 and Maximum Score: 10 Higher scores indicate worse outcomes.
Time Frame: up to 1 hour
Population: Nurse maximum pain score not documented for 2 subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
score on a scale
  15 minutes | 3.56 (3.45) | 2.47 (3.04)
  30 minutes | 2.28 (2.70) | 1.88 (2.67)
  Nurse Max Score up to 1 hour: number analyzed (Participants) | 17 | 16
  Nurse Max Score up to 1 hour | 5.29 (4.30) | 5.69 (4.27)

2. Secondary Outcome: Number of Participants With Nausea, Vomiting, Pruritis
Description: Collected in recovery room and asked in questionnaires, collected from parents on post-operative days 1, 5, and 30.
Time Frame: up to post-op day 30
Measure: Number; unit: participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
participants
  Nausea | 2 | 1
  Vomiting | 2 | 0
  pruritis | 0 | 0

3. Secondary Outcome: Number of Participants Who Sought Unplanned Medical Attention
Description: Number of participants who were readmitted to the hospital and sought unplanned medical attention (phone calls, office visits, emergency department visits) by chart review and questionnaires for readmission and medical reattendance, including calls to physician
Time Frame: up to post-op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
Participants | 1 | 3

4. Secondary Outcome: Number of Participants Who Were Readmitted to the the Hospital
Description: Number of participants who were readmitted to the hospital by chart review and questionnaires for readmission and medical reattendance, including calls to physician.
Time Frame: Up to post-op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
Participants | 1 | 0

5. Secondary Outcome: Number of Participants With Non-artefactual Percentage of Oxygen Saturation (SpO2)<90% (>30 Seconds)
Description: Number of participants with non-artefactual percentage of oxygen saturation (SpO2) less than 90% for greater than 30 seconds). Collected in the recovery room and chart review
Time Frame: up to post-op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
Participants | 1 | 1

6. Secondary Outcome: Number of Patients Receiving Rescue Opioids
Description: How many subjects received rescue opioids after surgery
Time Frame: up to post-op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
Participants | 9 | 11

7. Secondary Outcome: Family Satisfaction With Patient Recovery Based on Five-point Likert Score
Description: Follow-up questionnaire to family on post-op days 1, 5, and 30. Parents will be asked to rank how satisfied they are with their child's recovery by using these two prompts: "I am satisfied with my child's recovery," and "I am satisfied with my child's pain control at home." They will choose from the following options: "Strongly agree = 1", "Agree = 2", "Undecided = 3", "Disagree = 4", "Strongly Disagree =5." Minimum score is 1, Max is 5. Higher scores indicate worse outcomes. Data assessed at post-op days 1, 5, and 30 were averaged.
Time Frame: assessed at post-op days 1, 5, and 30
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
score on a scale
  Recovery Satisfaction | 1.4 [1 to 3] | 1.3 [1 to 3]
  Pain Control Satisfaction | 1.6 [1 to 4] | 1.5 [1 to 3]

8. Secondary Outcome: Number of Participants That Experienced Any Post-operative Bleeding Throughout the Study
Description: Follow-up questionnaires administered on post-operative day 1, 5, ad 30 and chart review.
  Question: Has your child had any bright red blood in their mouth? Answer options: Yes/No
Time Frame: up to post-op day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
Number analyzed (Participants) | 18 | 17
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days
Description: Definitions of adverse and/or serious adverse events do not differ from clinicaltrials.gov
Arm/Group | Traditional Care Group (TCG) | Opioid-Free Group (OFG)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/17
Other Adverse Events (participants affected / at risk) | 4/18 | 6/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Care Group (TCG) (N=18) | Opioid-Free Group (OFG) (N=17)
Prolonged admission (General disorders) | 1 (1) | 0 (0)
Readmission (General disorders) | 1 (1) | 0 (0)
Bleeding Events (Surgical and medical procedures) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Traditional Care Group (TCG) (N=18) | Opioid-Free Group (OFG) (N=17)
Oxygen Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dehydration (General disorders) | 1 (1) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Emergency department encounter (Surgical and medical procedures) | 1 (1) | 4 (4)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04528173/Prot_SAP_004.pdf
  • Informed Consent Form (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT04528173/ICF_005.pdf